CLINICAL TRIAL: NCT06520670
Title: Urinary galectin_3 Binding Protein as a Novel Biomarker in Lupus Nephritis and Indicator for Disease Activity
Brief Title: Urinary G3BP as a Novel Biomarker in Lupus Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Mahmoud Hussien Ali, Principal investigator, Assiut University
Other Study IDs: Urinary G3BP in LN
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with Lupus nephritis diagnosed by biopsy.
  Interventions: Diagnostic Test: Urinary galectin-3 binding protein
- Patient with SLE without nephritis.
  Interventions: Diagnostic Test: Urinary galectin-3 binding protein
- Patient with nephritis of other reasons: Patient with nephritis of other reasons; acute proliferative glomerulonephritis (postinfectious and infection associated), crescentic glomerulonephritis, else.
  Interventions: Diagnostic Test: Urinary galectin-3 binding protein

INTERVENTIONS:
Diagnostic Test: Urinary galectin-3 binding protein — Investigate urinary galectin-3 binding protein (G3BP) as a biomarker for lupus nephritis and indicator for disease activity.

SUMMARY:
Estimation of urinary Galectin-3 binding protein (u-Gal-3BP) in patients with systemic lupus erythematosus with and without lupus nephritis and in glomerulonephritis for other kidney diseases, Find the relation of urinary Galectin-3 binding protein (u-Gal-3BP) levels with lupus nephritis, and Correlate urinary Galectin-3 binding protein (u-Gal-3BP) levels with SLE disease activity

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a systemic autoimmune disease with multisystem involvement. The condition has several phenotypes, with varying clinical presentations from mild mucocutaneous manifestations to multiorgan and severe central nervous system involvement. Several immunopathogenic pathways play a role in the development of SLE. Hargraves described the lupus erythematosus (LE cell) in 1948. Several pathogenic autoantibodies have since been identified. Despite recent advances in technology and understanding of the pathological basis and risk factors for SLE, the exact pathogenesis is still not well known. Diagnosis of SLE can be challenging, and while several classification criteria have been posed, their utility in the clinical setting is still a matter of debate. Management of SLE is dictated by organ system involvement. Despite several agents shown to be efficacious in treating SLE, the disease still poses significant morbidity and mortality risk in patients.

Lupus nephritis (LN) is a highly prevalent and serious clinical manifestation among patients with systemic lupus erythematosus (SLE). It affects up to 60% of patients, depending on the examined cohort. Although SLE management has improved, LN still represents a difficult to treat manifestation, with renal flares occurring in about half of the patients and development of end stage renal disease (ESRD) in 5%20% of patients.

Lupus nephritis directly contributes to SLE-related mortality, both in the early and later disease phase.

Lupus nephritis diagnosis relies on kidney biopsy, which is instrumental for histological characterization, and treatment decisions. However, the biopsy procedure is invasive, often associated with discomfort for the patient, and sometimes with bleeding complications. Although repeated biopsies have been shown to be of value, their utility still remains controversial for verifying treatment effects, monitoring disease and predicting outcomes in clinical practice.

In this context, it is highly desirable to identify new non-invasive biomarkers that may reflect the type of kidney involvement, reflect the degree of histological activity and damage, predict LN flares and be useful for assessing treatment response. In this respect, urinary biomarkers are of high relevance since they can serve as liquid biopsy and reveal pathogenic events taking place in the kidney.

the investigators investigated urinary Galectin-3 binding protein (u-Gal-3BP) as a novel candidate biomarker for disease activity in renal lupus, here studied in a real life SLE cohort.

Gal-3BP is an interferon-inducible secreted scavenger protein belonging to the lectin family. in SLE, previous studies have demonstrated high expression of Gal-3BP in blood, both in systemic and cutaneous forms of lupus, and the protein was found in circulating macrovesicles, as well as in macrovesicles in the context of immune deposits in the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Any age above 18 years.
* Patient with Lupus nephritis diagnosed by biopsy.
* Patient with SLE without nephritis.
* Patient with nephritis of other reasons; acute proliferative glomerulonephritis (postinfectious and infection associated), crescentic glomerulonephritis, else.

Exclusion Criteria:

* Pregnant.
* Patient who refused to be part of the study.
* Patients with estimated Glomerular Filtration Rate less than 15ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: males and females that are not pregnant of any age above 18 years have one of next criteria:
  * Patient with Lupus nephritis diagnosed by biopsy.
  * Patient with SLE without nephritis.
  * Patient with nephritis of other reasons; acute proliferative glomerulonephritis (postinfectious and infection associated), crescentic glomerulonephritis, else.
  All patients were selected from outpatient clinic of rheumatology and inpatient wards of Internal Medicine Department Assiut University Hospitals. The patients will be interviewed, and those who agreed to share in the study were selected. An informed consent was obtained from each patient to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Level of galectin_3 binding protein in urine samples . | baseline
  Level of galectin_3binding protein in urine samples by pg/mmol using ELISA in patient with lupus nephritis.